CLINICAL TRIAL: NCT05646758
Title: A Phase I Clinical Trial Evaluating the Tolerance and Pharmacokinetics of TQB2934 for Injection in Multiple Myeloma Subjects
Brief Title: A Clinical Trial of TQB2934 for Injection in Multiple Myeloma Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2934-I-01
Record Dates: First submitted 2022-12-01; First posted 2022-12-12 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2934 injection (Experimental): intravenous injection. 0.09mg, 0.36 mg, 1mg, 2mg, 3mg, 5mg, 6mg, 10mg, 12mg, 16mg, 20mg each time.
  once a week in Cycle 1-3. once every 2 weeks in Cycle 4-6. if reach PR and above remission after 6 cycles of administration, once every 4 weeks,28 days as a treatment cycle.
  Interventions: Drug: TQB2934 injection

INTERVENTIONS:
Drug: TQB2934 injection — TQB2934 is an anti-CD3×BCMA double-specific antibody，which at one end binds to the CD3 receptor on the surface of T cells ,and the other end binds to BCMA to recruit T cells around BCMA-positive cells, which can activate T cells .Active T cells release granzyme and perforin to kill BCMA-positive target cells.

SUMMARY:
TQB2934 is an anti-CD3(Early T Cell Marker)×BCMA (B cell maturation antigen) double-specific antibody，and the isoform is IgG1 (Native Immunoglobulin G1), which at one end binds to the CD3 receptor on the surface of T cells ,and the other end binds to BCMA(B cell maturation antigen) to recruit T cells around BCMA-positive cells, which can activate T cells .Active T cells release granzyme and perforin to kill BCMA-positive target cells.TQB2934 for injection is planned for the treatment of patients with multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* The subjects volunteered to join the study and signed informed consent form (ICF)with good compliance;
* Age: ≥ 18 years old (when signing ICF); ECOG PS score: 0-1; The expected survival period is more than 3 months;
* Multiple myeloma with diagnostic records and meeting the IMWG diagnostic criteria;
* In the presence of measurable lesions, at least one of the following criteria must be met:

  1. Serum monoclonal immunoglobulin (M protein)≥1.0g/dL,or urine M protein≥200mg/24h;
  2. Light chain type: serum immunoglobulin free light chain (FLC) ≥ 10 mg/dL, and the ratio of free light chain serum immunoglobulin κ and λ is abnormal;
* Relapsed or refractory multiple myeloma who have received at least 1 line of therapy in the past, and are refractory to at least 1 proteasome inhibitor (PI), 1 immunomodulator (IMiD) and 1 CD38 monoclonal antibody;
* Disease progression during or within 12 months after the last treatment (meeting the PD criteria of IMWG), including refractory or no remission of the last treatment (≥1 cycle) or disease progression within 6 months;
* Major organ function is good;
* Female subjects of childbearing age should agree to use contraceptive measures (such as intrauterine devices, contraceptives or condoms) during the study period and within 6 months after the end of the study; serum pregnancy/urine pregnancy test within 7 days before study enrollment;

Exclusion Criteria:

* Comorbidities and medical history:

  1. Other malignant tumors have occurred or are currently suffering from other malignant tumors within 3 years before the first medication.
  2. Unresolved toxic reactions higher than CTC AE grade 1 or higher due to any previous treatment, excluding alopecia, fatigue and peripheral neuropathy;
  3. Major surgical intervention, open biopsy, or significant traumatic injury within 28 days prior to first dose;
  4. long-term unhealed wounds or fractures;
  5. Hyperactive/venous thrombosis events occurred within 6 months before the first medication, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc.;
  6. Those who have a history of psychotropic drug abuse and cannot quit or have mental disorders;
  7. Subjects with any severe and/or uncontrolled disease,include:

     1. Unsatisfactory blood pressure control (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg, at least 2 measurements at intervals of more than 24 hours);
     2. Myocardial infarction, unstable angina, CTC AE ≥ grade 2 stable angina, ≥ grade 2 heart failure (New York Heart Association (NYHA) classification), ≥ grade 2 arrhythmia occurred within 6 months before the first medication;
     3. Cardiac ultrasound evaluation: left ventricular ejection fraction (LVEF) <50%;
     4. Active or uncontrolled severe bacterial, viral or systemic fungal infection within 28 days before the first dose (≥CTC AE grade 2 infection);
     5. Hepatitis (meeting one of the following criteria: hepatitis B: HBV DNA detection value exceeds the upper limit of normal value; hepatitis C: HCV RNA detection value exceeds the upper limit of normal value) or decompensated cirrhosis (Child-Pugh grade B, C grade;
     6. Chronic obstructive pulmonary disease (COPD) and forced expiratory volume in 1 second (FEV1) <60% of predicted value.
     7. Has developed or currently suffered from asthma within 2 years before the first medication;
     8. A history of immunodeficiency, including HIV positive or other acquired, congenital immunodeficiency diseases, or a history of solid organ transplantation (except corneal transplantation), and active or autoimmune patients who need to receive systemic immunosuppressant therapy;
     9. Poorly controlled diabetes (fasting blood glucose (FBG) >10mmol/L);
     10. Suffering from epilepsy and needing treatment;
* Tumor-related symptoms and treatment:

  1. Diagnosed with amyloidosis, plasma cell leukemia (PCL, peripheral plasma cell ratio ≥ 20%, or absolute plasma cell count ≥ 2×109/L), Waldenstrom macroglobulinemia (WM) or POEMS syndrome;
  2. Known multiple myeloma meningeal or central nervous system invasion or highly suspected meningeal or central nervous system invasion but cannot be identified;
  3. Previously received BCMA-targeted therapy;
  4. Previously received allogeneic hematopoietic stem cell transplantation or chimeric antigen receptor T (CAR-T), CAR-NK cell therapy; or received autologous hematopoietic stem cell transplantation (ASCT) within 12 weeks before the first drug;
  5. Received targeted therapy, cytotoxic drugs or any antibody therapy within 3 weeks before the first medication; received proteasome inhibitor therapy or radiotherapy within 2 weeks before the first medication; received immunomodulator therapy within 1 week before the first medication.(Prophylaxis to prevent infusion-related reactions prior to study drug administration)(Calculate the washout period from the end of the last treatment);
* research treatment related:

  1. History of live attenuated vaccine vaccination within 28 days before the first dose or planned live attenuated live vaccine vaccination during the study;
  2. Unexplained severe allergy history, known allergy to monoclonal antibody drugs or exogenous human immunoglobulin, or known allergy to TQB2934 for injection or excipients in pharmaceutical preparations;
* Those who have participated in other anti-tumor drug clinical trials within 4 weeks before the first drug use or have not exceeded 5 drug half-lives;
* According to the investigator's judgment, there are concomitant diseases that seriously endanger the safety of the subjects or affect the completion of the study, or subjects who are considered unsuitable for enrollment for other reasons;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-03-17 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Up to 18 months
  DLT refers to any of the toxicity events in the first administration of TQB2934 for injection to the end of the first treatment cycle.
Maximum Tolerated Dose (MTD) | Up to 18 months
  After the trial, ordinal regression was used to determine the maximum tolerated dose (MTD)
Incidence and severity of serious adverse events (AEs) | Up to 18 months
  Incidence and severity of serios adverse events (AEs) will be reported for safety evaluation.
Incidence and severity of adverse events (AEs) | Up to 18 months
  Incidence and severity of adverse events (AEs) will be reported for safety evaluation.
Incidence and severity abnormal laboratory test value | Up to 18 months
  Incidence and severity abnormal laboratory test value will be reported for safety evaluation.

SECONDARY OUTCOMES:
Elimination half-life (t1/2) | 120 hours after administration
  t1/2 is time it takes for the blood concentration of TQB2934 to drop by half.
Area under the plasma concentration-time curve (AUC0-last) | 120 hours after administration
  To characterize the pharmacokinetics of TQB2934 by assessment of area under the plasma concentration time curve.
Apparent clearance (CL) | 120 hours after administration
  Apparent clearance (CL) after administration
Terminal phase apparent volume of distribution (Vz) | 120 hours after administration
  Terminal phase apparent volume of distribution (Vz)
Plasma trough concentration (Cmin) | 120 hours after administration
  Cmin is the minimum plasma concentration of TQB2934.
Overall response rate (ORR) | Up to 18 months
  Proportion of subjects with best response as PR(Partial relief), VGPR(Very good partial relief), CR(Complete Response), sCR(Strict Complete Response)
Clinical benefit rate (CBR) | Up to 18 months
  Proportion of subjects with best response as MR(Minor relief), PR(Partial relief), VGPR(Very good partial relief), CR(Complete Response), sCR(Strict Complete Response)
Very good partial response rate (VGPR) | Up to 18 months
  Proportion of subjects whose best response is VGPR, CR, sCR;
Complete Response (CR) / Strict Complete Response (sCR) Rate | Up to 18 months
  Proportion of subjects whose best response is CR and sCR;
Negative rate of minimal residual disease (MRD) | Up to 18 months
  The proportion of subjects with negative MRD (<10-5, multicolor flow cytometry or next-generation sequencing) at any time point from the first administration of the trial drug to disease progression or before receiving new anti-tumor therapy;
Duration of remission (DOR) | Up to 18 months
  For all subjects whose best response was PR, VGPR, CR, sCR, the time from the date of first achieving PR, VGPR, CR, sCR to the date of first definite disease progression or (any cause) death(whichever occurs first).
Time to first remission (TTR) | Up to 18 months
  Among all the subjects whose best response is PR, VGPR, CR, sCR, the time from the first administration of the test drug to the date of the first PR and above remission.
Progression-free survival (PFS) | Up to 18 months
  The time between the first dose of the trial drug and the date of first definite disease progression or death (from any cause), whichever occurs first.
Overall survival (OS) | Up to 18 months
  Time from first dose of study drug to date of death from any cause.
Disease status was determined using the International Myeloma Working Group (IMWG) 2016 criteria | Up to 18 months
  Disease status was determined using the International Myeloma Working Group (IMWG) 2016 criteria
Antidrug antibody (ADA) incidence | Up to 18 months
  Positive incidence of anti-drug antibodies
Peripheral blood soluble BCMA (sBCMA) level | Up to 18 months
  The level of soluble BCMA (sBCMA) in peripheral blood is the pharmacodynamic index of TQB2934.
Receptor occupancy rate (RO) | Up to 18 months
  The receptor occupation (RO) of TQB2934 on immune cells in human body
Cytokine Interleukin 2 (IL-2) levels | Up to 18 months
  The level of cytokine interleukin 2 (IL-2) is the pharmacodynamic index of TQB2934.
Cytokine Interleukin 6 (IL-6) levels | Up to 18 months
  The level of cytokine interleukin 6 (IL-6) is the pharmacodynamic index of TQB2934.
Cytokine Interleukin 10 (IL-10) levels | Up to 18 months
  The level of cytokine interleukin 10 (IL-10) is the pharmacodynamic index of TQB2934.
Cytokine Interferon γ (IFN-γ) levels | Up to 18 months
  The level of cytokine Interferon γ (IFN-γ) is the pharmacodynamic index of TQB2934.
Cytokine Interferon α (IFN-α) levels | Up to 18 months
  The level of cytokine Interferon α (IFN-α) is the pharmacodynamic index of TQB2934.

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Sun Yat-Sen University Cancer Canter, Guangzhou, Guangdong
  - The Henan Cancer Hospital, Zhengzhou, Henan
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Shandong First Medical University Affiliated Tumor Hospital, Jinan, Shandong
  - Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No